CLINICAL TRIAL: NCT05298475
Title: Short-term Effect of Modified 、Low-dose Proprotein Convertase Subtilisin/Kexin Type 9 Inhibitor Combined With Stains on Serum Lipids in Chinese Population With Acute Coronary Syndrome : the Singe-center 、Real-world Study
Brief Title: Low-dose PCSK9 Inhibitor Combined With Stains on Serum Lipids in Chinese Population With Acute Coronary Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPICS-CHACS
Record Dates: First submitted 2022-03-13; First posted 2022-03-28 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute coronary syndrome; Serum lipids; PCSK9 inhibitor; Statin
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Statin-only group (Experimental): The patients in this group are treated with medium-dose statin daily(atorvastatin 20mg qn or rosuvastatin 10mg qn).
  Interventions: Drug: Statin
- Low-dose PCSK9 inhibitor group (Experimental): The patients in this group are treated with medium-dose statin daily(atorvastatin 20mg qn or rosuvastatin 10mg qn) and 1 injection of PCSK9 inhibitor once a month SC.
  Interventions: Drug: Statin; Drug: PCSK9 inhibitor
- Normal-dose PCSK9 inhibitor group (Experimental): The patients in this group are treated with medium-dose statin daily(atorvastatin 20mg qn or rosuvastatin 10mg qn) and 1 injection of PCSK9 inhibitor twice a month SC.
  Interventions: Drug: Statin; Drug: PCSK9 inhibitor

INTERVENTIONS:
Drug: Statin — Medium-dose statin daily(atorvastatin 20mg qn or rosuvastatin 10mg qn)
Drug: PCSK9 inhibitor — 1 injection of PCSK9 inhibitor once a month SC
  Arms: Low-dose PCSK9 inhibitor group
Drug: PCSK9 inhibitor — 1 injection of PCSK9 inhibitor twice a month SC
  Arms: Normal-dose PCSK9 inhibitor group

SUMMARY:
A total of 100 patients aged 18-85 years old with a definite diagnosis of ACS were admitted to the Department of Cardiovascular, The First Affiliated Hospital of Nanjing Medical University. These patients had fasting serum low-density lipoprotein (LDL-C) >1.8mmol/L (70mg/dL) and were divided into three groups according to the lipid-lowering regimen used: a total of 50 people in the statin-only group received a daily oral medium-dose statin (atorvastatin 20mg qn or rosuvastatin 10mg qn); a total of 30 people in the statin + one injection group per month received oral atorvastatin 20mg qn or rosuvastatin 10mg qn + once a month, subcutaneous injection of 1 injection of PCSK9 inhibitor each time; the remaining 20 people were divided into statin + two injections per month group, oral atorvastatin 20mg qn or rosuvastatin 10mg qn + twice a month, subcutaneous injection of 1 injection of PCSK9 inhibitor each time. We followed up the blood lipid levels of these patients at different time points (one month,three month, six month), including TC, TG, HDL-C, LDL-C,taking the LDL-C reduction ≥50% from the baseline, LDL-C<1.8mmol/L (70mg/dL), and LDL-C<1.4mmol/L (55mg/dL) as the the compliance standard, the blood lipid compliance rates of the three groups at the 6th month of treatment were calculated respectively. The adverse drug reactions of the patients during follow-up were recorded.

DETAILED DESCRIPTION:
Purpose:The purpose of this study was to explore the short-term effect of a modified, lower-than-guideline-recommended doses of PCSK9 inhibitors combined with a statin in the treatment of dyslipidemia in Chinese with the acute coronary syndrome (ACS), to provide evidence for the use of this drug in real-world Chinese populations. This study will provide more economical, convenient, and acceptable treatment options.

A total of 100 patients aged 18-85 years old with a definite diagnosis of ACS were admitted to the Department of Cardiovascular, The First Affiliated Hospital of Nanjing Medical University. These patients had fasting serum low-density lipoprotein (LDL-C) >1.8mmol/L (70mg/dL) and were divided into three groups according to the lipid-lowering regimen used: a total of 50 people in the statin-only group received a daily oral medium-dose statin (atorvastatin 20mg qn or rosuvastatin 10mg qn); a total of 30 people in the statin + one injection group per month received oral atorvastatin 20mg qn or rosuvastatin 10mg qn + once a month, subcutaneous injection of 1 injection of PCSK9 inhibitor each time; the remaining 20 people were divided into statin + two injections per month group, oral atorvastatin 20mg qn or rosuvastatin 10mg qn + twice a month, subcutaneous injection of 1 injection of PCSK9 inhibitor each time. We followed up the blood lipid levels of these patients at different time points (one month,three month, six month), including TC, TG, HDL-C, LDL-C, taking the LDL-C reduction ≥50% from the baseline, LDL-C<1.8mmol/L (70mg/dL), and LDL-C<1.4mmol/L (55mg/dL) as the the compliance standard, the blood lipid compliance rates of the three groups at the 6th month of treatment were calculated respectively. The adverse drug reactions of the patients during follow-up were recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-85 years, gender unlimited;
2. Diagnosed with acute coronary syndrome;
3. The fasting LDL-C≥1.8mmol/L (70mg/dL);
4. Subjects participated in the study voluntarily and signed informed consent.

Exclusion Criteria:

1. Uncontrolled hypertension defined as sitting systolic blood pressure (SBP) > 180 mmHg or diastolic BP (DBP) > 110 mmHg；
2. Last known left ventricular ejection fraction < 30%
3. Known hemorrhagic stroke at any time；
4. Severe renal dysfunction, defined as an estimated glomerular filtration rate (eGFR) < 20 mL/min/1.73m2 at final screening；
5. Active liver disease or hepatic dysfunction, defined as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 times；
6. LDL or plasma apheresis within 12 months prior to randomization；
7. Pregnant or lactating women；
8. Severe, concomitant non-cardiovascular disease that is expected to reduce life expectancy to less than 3 years；
9. Patients allergic to PCSK9 inhibitors.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
The level of total cholesterol(TC) | 6 month
  The level of total cholesterol(TC) at 6 month
The level of triglyceride(TG) | 6 month
  The level of triglyceride(TG) at 6 month
The level of high-density lipoprotein cholesterol(HDL-C) | 6 month
  The level of high-density lipoprotein cholesterol(HDL-C) at 6 month
The level of low-density lipoprotein cholesterol(LDL-C) | 6 month
  The level of low-density lipoprotein cholesterol(LDL-C) at 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China